CLINICAL TRIAL: NCT05051306
Title: Effects of Volume-matched Resistance Exercise With Different Loads on Metabolic Responses
Brief Title: Effects of Resistance Exercise on Metabolic Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 202011HM005
Record Dates: First submitted 2021-08-30; First posted 2021-09-21 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Inflammatory Response
Keywords: resistance exercise; equal training volume; immune response

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-load resistance exercise (Experimental): 4 high-load resistance exercises that target all major muscle groups.
  Interventions: Other: High-load resistance exercise
- Low-load resistance exercise (Experimental): 4 low-load resistance exercises that target all major muscle groups.
  Interventions: Other: Low-load resistance exercise
- Sedentary control (No Intervention): Subjects in control trial stayed sedentary during the period.

INTERVENTIONS:
Other: High-load resistance exercise — Subjects in high-load trial performed 4 sets per exercise, 8 repetitions with load of 85%-8RM with 90 sec of rest between sets.
  Arms: High-load resistance exercise
Other: Low-load resistance exercise — Subjects in low-load trial performed 4 sets per exercise, 15 repetitions with load of 45%-8RM with 90 sec of rest between sets.
  Arms: Low-load resistance exercise

SUMMARY:
Healthy young adults will complete three trials in a randomized crossover counter-balanced order, including two different loads of resistance exercise and sedentary control. During each trial, blood samples will be collected.

The investigators hypothesized that high-load and low-load resistance exercise exert similar metabolic responses.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-30
* Healthy male
* Without experience of resistance training

Exclusion Criteria:

* No acute or chronic musculoskeletal symptoms
* Smoking
* Alcohol or drug abuse
* Fail to conduct resistance exercise

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 11 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-03-07 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in glucose | 4-hour during each study intervention
  glucose in mg/dL
Changes in insulin | 4-hour during each study intervention
  insulin in mU/L
Changes in TG | 4-hour during each study intervention
  TG mg/dL
Changes in uric acid | 4-hour during each study intervention
  uric acid mg/dL.

SECONDARY OUTCOMES:
Changes in biomarkers of inflammation | 4-hour during each study intervention
  Biomarkers of inflammation will be measured such as IL-10 in pg/mL and IL-6 in pg/mL.
Changes in cortisol | 4-hour during each study intervention
  cortisol in ng/mL
Changes in lactate | 4-hour during each study intervention
  lactate in mmol/L
Changes in complete blood count | 4-hour during each study intervention
  blood cell count in count per µL
Borgs Ratings of Perceived Exertion (RPE) | 1-hour during each exercise intervention
  Borgs RPE is a method of estimating exertion rating, based on a 6 to 20 rating scale (6 being the no exertion at all, 20 being maximal exertion).
Changes in ET-1 | 4-hour during each study intervention
  ET-1 in pg/mL
Changes in NO | 4-hour during each study intervention
  NO in µmol/L
Changes in biomarkers of muscle damage | 4-hour during each study intervention
  Biomarkers of muscle damage will be measured such as CK in U/L and LDH in U/L.
Heart rate (HR) | 6-hour during each study intervention
  HR will be measured during each study intervention.
Visual Analogue Scale (VAS) of appetite | 6-hour during each study intervention
  Hunger, fullness, desire to eat, and prospective food consumption will be measured via VAS ratings, based on a 100 mm long scale (0 being "not at all", 100 being "extremely").
Changes in biomarkers of appetite | 4-hour during each study intervention
  Biomarkers of appetite will be measured such as ghrelin in pg/mL and PYY in pg/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Wen Liu, Ph.D., Principal Investigator — National Taiwan Normal University
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No